CLINICAL TRIAL: NCT01561976
Title: The Effect of Food on the Pharmacokinetics of Metformin Given Either as Metformin Hydrochloride SR 1000mg Tablet or as a Fixed Dose Combination of Metformin Hydrochloride SR 1000mg/Glimepiride 2mg Tablet in Healthy Indian Volunteers.
Brief Title: Evaluation of Food Effect on the Pharmacokinetics of Sustained Release Metformin in Healthy Indian Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116519
Record Dates: First submitted 2012-02-16; First posted 2012-03-23 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin hydrochloride prolonged release (Active Comparator): 1000mg in fasting state
  Interventions: Drug: Metformin hydrochloride prolonged release
- metformin hydrochloride prolonged release (Active Comparator): 1000mg In fed state
  Interventions: Drug: metformin hydrochloride prolonged release
- Metformin hydrochloride sustained release/Glimepiride (Active Comparator): 1000/2mg In fed state
  Interventions: Drug: Metformin hydrochloride sustained release/Glimepiride

INTERVENTIONS:
Drug: Metformin hydrochloride prolonged release — 1000mg in fasting state
  Arms: Metformin hydrochloride prolonged release
Drug: metformin hydrochloride prolonged release — 1000mg in fed state
  Arms: metformin hydrochloride prolonged release
Drug: Metformin hydrochloride sustained release/Glimepiride — 1000/2mg in fed state
  Arms: Metformin hydrochloride sustained release/Glimepiride

SUMMARY:
Metformin hydrochloride in its immediate release (IR) form has been successfully used for decades in the treatment of type 2 diabetes; however the IR formulation may be associated with gastrointestinal side effects (especially nausea, diarrhea) in 20-30% patients, which can limit the tolerated dose, reduce adherence and result in discontinuation of therapy. Metformin hydrochloride extended release formulations have been developed to overcome these problems. In India, extended release formulations of metformin hydrochloride include metformin SR 1000mg tablet and combination of metformin hydrochloride SR 1000mg/glimepiride 2mg tablet. In the combination tablet, only metformin hydrochloride is in the extended release form. In view of the fact that extended release metformin hydrochloride is usually recommended with a meal, that food is known to affect the pharmacokinetic (PK) parameters of metformin and that there is a potential for dose dumping with extended release formulations that may lead to side effects similar to IR formulations, a study to estimate the magnitude of the food effect for these formulations in fed state compared to the fasting state is warranted. This study will be a randomized, single-center, open-label, single-dose, three-period, 6 sequence crossover study in 30 healthy adult volunteers to estimate the bioavailability of metformin from metformin hydrochloride 1000mg SR tablet given in fasting condition relative to metformin hydrochloride 1000mg SR tablet and a fixed dose combination of metformin hydrochloride 1000mg SR /glimepiride 2mg tablet, each given in fed condition. The safety and tolerability profile of metformin SR 1000mg tablet and metformin hydrochloride SR 1000mg/glimepiride 2mg tablet will also be evaluated in this study. The primary PK endpoints will be Cmax and AUC (0-∞). The secondary PK endpoints will include AUC (0-t), Tmax , T lag, Kel and t1/2. Safety endpoints will include vital signs, ECG, physical examination, clinical laboratory tests and adverse event reporting.

DETAILED DESCRIPTION:
Background:

Metformin hydrochloride, a biguanide, is an effective treatment for type 2 diabetes, lowering both basal and postprandial hyperglycemia either as monotherapy or in combination with other antihyperglycemic drugs. Metformin hydrochloride in its immediate release form (IR) has been used for decades in the treatment of type 2 diabetes. An IR formulation releases the entire drug within 1-2 h after dosing, resulting in high drug concentrations in the GI (gastrointestinal) tract which may be associated with GI side effects (especially nausea, diarrhea) in 20-30% patients. This can limit the tolerated dose, reduce adherence and result in discontinuation of therapy. In addition, the frequent need to administer metformin two or three times daily may also not support good adherence to therapy.

Metformin hydrochloride extended release (ER) formulations have been developed to overcome these problems. Because metformin gets absorbed in the first part of the small intestine, extended release metformin hydrochloride formulations employ various novel gastric-retentive techniques. The polymeric matrix (hydroxyl propyl methyl cellulose) of the extended release metformin tablet is designed to swell in the gastric fluid. As the matrix swells, it becomes resistant to peristalsis and is more easily retained in the stomach. Gastric fluid penetrates the matrix, dissolving the drug which then diffuses out of the matrix in the liquefied form. Metformin hydrochloride is thus slowly released from the matrix of the tablet and is absorbed when this gastric fluid passes through the small intestine. The slow release of the drug in the GI tract permits once daily dosing and also reduces the incidence of nausea (6.5%) and diarrhea (9.6%). These factors are particularly relevant for increasing treatment adherence to long term therapies like anti-diabetic medication.

Glimepiride, a new generation sulphonylurea, in doses of 1-8mg/day, is an effective treatment option for non-insulin dependent diabetes mellitus (NIDDM) patients. Oral bioavailability is approximately 100% and the absence of a food interaction guarantees highly reproducible pharmacokinetics with this drug. A combination tablet formulation of sustained release metformin hydrochloride and glimepiride is beneficial in terms of convenience of administration and patient compliance.

Metformin hydrochloride extended-release formulation should generally be given once daily with the evening meal. Administration with food increases the bioavailability of metformin hydrochloride. Food increases the extent of absorption (AUC) of metformin hydrochloride (AUC 13306 ng h/ml with high fat breakfast, AUC 10200 ng h/ml with a low fat breakfast, AUC 7506 ng h/ml in fasting condition). Food can either cause no change or an increase in Cmax of the drug. One study has reported no effect of food on the Cmax of metformin [high fat meal (1018 ng/ml), low fat meal (992 ng/ml) and fasting condition (1022 ng/ml)]. In contrast, in a healthy volunteer study with Glucophage SR 1000mg, food increased the extent of absorption (AUC) by 77%, peak plasma concentration (Cmax) by 26% and prolonged time to peak plasma concentration (Tmax) by about 1 hour as compared to the fasting state.

The mechanical stress of the grinding action of the stomach in the fed state could introduce variability if an extended release tablet containing metformin hydrochloride is broken down more rapidly than anticipated. Because food prolongs the gastric retention time, extended release formulations administered with food are exposed to longer duration of mechanical stress in the stomach. The latter raises the possibility of increased release rate (than intended) of the drug from the formulation. This can result in a higher risk of 'dose dumping', creating a potential safety risk for patients. Therefore it is clinically important to assess the effect of food on extended release formulations of metformin hydrochloride and metformin hydrochloride/glimepiride.

Study Rationale:

Extended release formulations of metformin hydrochloride in India include metformin SR 1000mg tablet and metformin hydrochloride SR 1000mg/glimepiride 2mg tablet. In the combination tablet, only metformin hydrochloride is in the extended release form. In view of the fact that extended release metformin hydrochloride is usually recommended with a meal, that food is known to affect the PK parameters of metformin and that there is a potential for dose dumping with extended release formulations that may lead to side effects similar to IR formulations, a study to estimate the magnitude of the food effect for these formulations in fed state compared to the fasting state is warranted. The safety and tolerability profile of metformin SR 1000mg tablet and metformin hydrochloride SR 1000mg/glimepiride 2mg tablet will also be evaluated in this study.

Objectives:

Primary:

To compare the pharmacokinetics and bioavailability of metformin given in a fed condition either as metformin hydrochloride 1000mg SR tablet or as a fixed dose combination of metformin hydrochloride 1000mg SR/glimepiride 2mg tablet with that given in fasting condition as metformin hydrochloride 1000mg SR tablet in healthy Indian volunteers.

Secondary:

To compare the safety and tolerability of metformin hydrochloride given in a fed condition either as metformin hydrochloride 1000mg SR tablet or as a fixed dose combination of metformin hydrochloride 1000mg SR/glimepiride 2mg tablet with that given in fasting condition as metformin hydrochloride 1000mg SR tablet in healthy Indian volunteers.

Study Design/Schematic:

This study will be a randomized, single-center, open-label, single-dose, three-period, 6 sequence crossover study in healthy adult volunteers to estimate the bioavailability of metformin from metformin hydrochloride 1000mg SR tablet given in fasting condition relative to metformin hydrochloride 1000mg SR tablet and a fixed dose combination of metformin hydrochloride 1000mg SR /glimepiride 2mg tablet, each given in fed condition.

30 healthy adult males will be randomized to receive a single dose of metformin hydrochloride SR (1000mg) in fasting state or metformin hydrochloride SR (1000mg) in fed state or a fixed dose combination of metformin hydrochloride 1000mg SR /glimepiride 2mg tablet in fed state in each treatment period. There will be 6 treatment sequences and a washout of 7 days between each of the three treatment periods.

Subjects will have a screening visit within 21 days prior to the first dose of study drug, followed by three treatment periods, each containing a single dose of study drug, followed by 30 hours of serial PK sample collection. Subjects will check out of the unit on Day +1 after collection of the 30 hour PK sample. Subjects will be instructed to return for the next treatment period or for the final follow-up visit, as appropriate. The final follow-up visit will occur 7 days after the last dose of study drug. Subjects will be assigned to each of the three treatments randomly as per the randomization schedule.

Study participants will check into the study unit of the clinical research organisation at least 12 hours prior to dosing and will remain in the clinical research unit up to 36 hours after the administration of the investigational product. In the fasting and fed conditions, the pre-dose dinner will be administered 11 hours prior to dosing of the drug.

Following a 10-hour overnight fast, subjects will be randomized as per predetermined randomization sequences to any of three study treatment arms in a ratio of 1:1:1 and then administered a single oral dose of study drug (A: metformin SR 1000 mg in fasting state, B: metformin SR 1000 mg in fed state, C: metformin SR 1000 mg/glimepiride 2 mg in fed state) in treatment period 1. In the subsequent two study periods, subjects will receive the other treatments, according to the randomisation schedule so that all subjects receive all treatments.

In the fasting condition, the dosing of the drug will take place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post dose respectively. On D+1 (day after the dosing day), breakfast and lunch will be provided at 25 hours and 30 hours post dose respectively.

In the fed condition, breakfast will be served at the scheduled time. The dosing of drug will be at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner will be served at 4, 9 and 13 hours post dose respectively. On D+1, breakfast and lunch will be provided at 25 hours and 30 hours post dose respectively.

According to CDSCO recommendations for high-fat breakfast for BA/BE fed state studies, participants must consume the high-fat breakfast (950-1000 kcal, at least 50% of calories from fat, 15-20% from protein and the rest from carbohydrates) approximately 15minutes prior to dosing. A random high fat breakfast sample served in the study will be sent for analysis and the caloric breakdown of the test meal will be calculated. In both, fasting and fed conditions, the study medication will be administered with 240 ml of a 20% glucose solution. Thereafter, 60 ml of a 20% glucose solution will be administered every 15 minutes for up to 4 hours after dosing.

In each period, a total of 18 blood samples will be collected using pre-labelled 6ml K3EDTA vacutainers as per the following schedule: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing. The volunteers will be housed for 36 hours after dosing. The bioanalyst will be blinded to study treatments received by the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, 12 lead ECG and chest-x-ray. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Medical Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Males between 18 and 50 years of age (both inclusive), who are willing to participate in the study and provide a written signed and dated informed consent.
3. Body weight more than or equal to 60 kg and BMI within the range 18.5-24.9 kg/m2 (inclusive).
4. Availability of a study volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

1. A positive pre-study urine drug screen.
2. A positive test for HIV antibody.
3. Subject has clinically significant abnormal values of laboratory parameters.
4. Regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits (CTRI, 2010).
5. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
6. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
7. Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator contraindicates their participation.
9. Where participation in another study would result in donation of blood or blood products in excess of 350 ml within a 90 day period prior to this study.
10. Unwillingness or inability to follow the procedures outlined in the protocol.
11. Subject is mentally or legally incapacitated or the subject is incapable of understanding the informed consent.
12. Subject has any evidence of impaired renal, hepatic, cardiac, lung or gastrointestinal function. Study volunteers with a history of tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for the study.
13. History of sensitivity to heparin or heparin-induced thrombocytopenia.
14. Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
15. Subject is intolerant to venipuncture.
16. Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2012-02-21 (Actual); Study Completion 2012-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] LIESEL DSILVA, JONATHAN PALMER, VISHWANATH SUDERSHAN, SANMAN GHORPADE, SADHNA JOGLEKAR . Effect of food on the absorption of metformin from sustained release metformin hydrochloride formulations in healthy Indian volunteers. Asian J Pharmaceut Clin Res. 2013;6(1):95-99.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one center in India from 30 January 2012 to 21 February 2012.
Pre-assignment Details: A total of 30 participants were enrolled in this study. METLEAD™ Forte SR (metformin hydrochloride prolonged release) and METLEAD™ G2 Forte (metformin hydrochloride sustained release/glimepiride) are registered product of GlaxoSmithKline.
Groups:
- METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting: In this sequence participants received single oral dose of METLEAD G2 Forte 1000 milligrams (mg)/2 mg tablet in fed state in period 1, METLEAD ForteSR 1000 mg tablet in fed state in period 2 and METLEAD ForteSR 1000 mg tablet in fasting state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1 (day after the dosing day), breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. Dosing was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post dose respectively.
- METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte: In this sequence participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fasting state in period 1, METLEAD ForteSR 1000 mg tablet in fed state in period 2 and METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. The dosing of drug was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting: In this sequence participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fed state in period 1, METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 2 and METLEAD ForteSR 1000 mg tablet in fasting state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. The dosing of drug was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed: In this sequence participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fasting state in period 1, METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 2 and METLEAD ForteSR 1000 mg tablet in fed state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. The dosing of drug was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte: In this sequence participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fed state in period 1, METLEAD ForteSR 1000 mg tablet in fasting state in period 2 and METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. The dosing of drug was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed: In this sequence participants received single oral dose of METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 1, METLEAD ForteSR 1000 mg tablet in fasting state in period 2 and METLEAD ForteSR 1000 mg tablet in fed state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. The dosing of drug was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
Period: Period 1
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed
Started | 5 | 5 | 4 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed
Started | 5 | 5 | 4 | 4 | 5 | 4
Completed | 5 | 5 | 4 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed
Started | 5 | 5 | 4 | 4 | 5 | 4
Completed | 4 | 5 | 3 | 4 | 5 | 4
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed
Started | 4 | 5 | 3 | 4 | 5 | 4
Completed | 4 | 5 | 3 | 4 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting: In this sequence participants received single oral dose of METLEAD G2 Forte 1000 mg/2 mg tablet in fed state in period 1, METLEAD ForteSR 1000 mg tablet in fed state in period 2 and METLEAD ForteSR 1000 mg tablet in fasting state in period 3. There was a washout period of 7 days between each treatment period. In the fasting and fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively. In the fed condition, breakfast was served at the scheduled time. Dosing was at the same scheduled time as dosing in the fasting condition. Lunch, snack and dinner was served at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- Total: Total of all reporting groups
Arm/Group | METLEAD G2 Forte, METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed, METLEAD G2 Forte | METLEAD ForteSR-Fed, METLEAD G2 Forte, METLEAD ForteSR-Fasting | METLEAD ForteSR-Fasting, METLEAD G2 Forte, METLEAD ForteSR-Fed | METLEAD ForteSR-Fed, METLEAD ForteSR-Fasting, METLEAD G2 Forte | METLEAD G2 Forte, METLEAD ForteSR-Fasting, METLEAD ForteSR-Fed | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.2 (5.63) | 25.6 (4.72) | 27.0 (5.79) | 31.8 (9.31) | 34.6 (6.73) | 25.4 (3.78) | 28.8 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 5 | 5 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  India | 5 | 5 | 5 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax)
Description: Pharmacokinetic (PK) blood samples for estimation of Cmax were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population included participants who received study medication. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Groups:
- METLEAD ForteSR-Fasting: Participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fasting state. In the fasting conditions, the pre-dose dinner was administered 11 hours prior to dosing. In fasting condition, dosing took place at the scheduled time followed by breakfast, lunch and dinner at 4, 8 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD ForteSR-Fed: Participants received single oral dose of METLEAD ForteSR 1000 mg tablet in fed state. In the fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In the fed condition, breakfast was served at the scheduled time. The dosing of drug took place at the scheduled time followed by lunch, snack and dinner at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
- METLEAD G2 Forte: Participants received single oral dose of METLEAD G2 Forte 1000 mg/2 mg tablet in fed state. In the fed conditions, the pre-dose dinner was administered 11 hours prior to dosing. In the fed condition, breakfast was served at the scheduled time. The dosing of drug took place at the scheduled time followed by lunch, snack and dinner at 4, 9 and 13 hours post-dose respectively. On D+1, breakfast and lunch was provided at 25 hours and 30 hours post-dose respectively.
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Nanograms per milliliter (ng/mL) | 884.297 (28.10) | 963.384 (26.13) | 942.653 (27.16)
Statistical Analysis 1: Comparison: METLEAD ForteSR-Fasting vs METLEAD ForteSR-Fed; Test type: Other; p = 0.1413, ANOVA; Ratio = 108.94, 95% CI 2-sided [101.01 to 117.50] — Ratio= METLEAD ForteSR-Fed/METLEAD ForteSR-Fasting
Statistical Analysis 2: Comparison: METLEAD ForteSR-Fasting vs METLEAD G2 Forte; Test type: Other; p = 0.1413, ANOVA; Ratio = 107.24, 95% CI 2-sided [99.37 to 115.73] — Ratio= METLEAD G2 Forte/METLEAD ForteSR-Fasting

2. Primary Outcome: Area Under Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time [AUC (0-infinity)]
Description: PK blood samples for estimation of AUC (0-infinity) were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms hour per milliliter (µ.hr/mL)
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Micrograms hour per milliliter (µ.hr/mL) | 10099.285 (30.31) | 11765.202 (24.99) | 10751.895 (29.76)
Statistical Analysis 1: Comparison: METLEAD ForteSR-Fasting vs METLEAD ForteSR-Fed; Test type: Other; p = 0.0171, ANOVA; Ratio = 116.50, 95% CI 2-sided [106.91 to 126.95] — Ratio= METLEAD ForteSR-Fed/METLEAD ForteSR-Fasting
Statistical Analysis 2: Comparison: METLEAD ForteSR-Fasting vs METLEAD G2 Forte; Test type: Other; p = 0.0171, ANOVA; Ratio = 107.24, 95% CI 2-sided [98.35 to 116.94] — Ratio= METLEAD G2 Forte/METLEAD ForteSR-Fasting

3. Secondary Outcome: AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments [AUC (0-t)]
Description: PK blood samples for estimation of AUC (0-t) were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µ.hr/mL
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
µ.hr/mL | 9894.580 (30.48) | 11563.589 (25.02) | 10546.905 (29.87)
Statistical Analysis 1: Comparison: METLEAD ForteSR-Fasting vs METLEAD ForteSR-Fed; Test type: Other; p = 0.0169, ANOVA; Ratio = 116.87, 95% CI 2-sided [107.07 to 127.57] — Ratio= METLEAD ForteSR-Fed/METLEAD ForteSR-Fasting
Statistical Analysis 2: Comparison: METLEAD ForteSR-Fasting vs METLEAD G2 Forte; Test type: Other; p = 0.0169, ANOVA; Ratio = 107.38, 95% CI 2-sided [98.30 to 117.29] — Ratio= METLEAD G2 Forte/METLEAD ForteSR-Fasting

4. Secondary Outcome: Time of Occurrence of Cmax (Tmax)
Description: PK blood samples for estimation of Tmax were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Hour | 8.00 [1.00 to 12.00] | 8.00 [4.50 to 12.00] | 8.00 [4.50 to 12.00]

5. Secondary Outcome: PK Lag Time (Tlag)
Description: PK blood samples for estimation of Tlag were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Hour | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.52] | 0.50 [0.00 to 0.52]

6. Secondary Outcome: Elimination Constant (Kel)
Description: PK blood samples for estimation of Kel were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Fraction/hour
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Fraction/hour | 0.162 [0.088 to 0.192] | 0.167 [0.144 to 0.209] | 0.165 [0.135 to 0.192]

7. Secondary Outcome: Terminal Phase Half Life (t1/2)
Description: PK blood samples for estimation of t1/2 were collected at 0.0 (pre-dose) and 0.5,1,2,2.5,3,3.5,4,4.5,5,6,7,8,10, 12, 16,24 and 30 hours after dosing. Point estimates and corresponding 90% confidence interval was constructed for the ratio of the geometric mean of the test treatment (fed condition) to the geometric mean of the reference treatment (fasting condition).
Time Frame: 0.0 (pre-dose) and 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24 and 30 hours after dosing
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Hour | 4.281 [3.604 to 7.915] | 4.155 [3.321 to 4.804] | 4.199 [3.610 to 5.153]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A serious adverse event is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect, medically significant or possible drug-induced liver injury.
Time Frame: Up to approximately 24 days (during treatment and washout) after initiation of study
Population: PK Population.
Measure: Count of Participants; unit: Participants
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
Number analyzed (Participants) | 24 | 24 | 24
Participants
  Any AEs | 0 | 1 | 2
  Any SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 24 days (during treatment and washout) after initiation of study. On treatment SAEs and non-serious AEs have been presented.
Description: PK population was used for the analysis of safety data.
Arm/Group | METLEAD ForteSR-Fasting | METLEAD ForteSR-Fed | METLEAD G2 Forte
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | METLEAD ForteSR-Fasting (N=24) | METLEAD ForteSR-Fed (N=24) | METLEAD G2 Forte (N=24)
Fever (General disorders) | 0 | 0 | 1
Upper abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Loose motions (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.